CLINICAL TRIAL: NCT07118904
Title: The Effect of Acute Dehydration on Sleep Quality, Cognitive Skills, and Electromyographic Responses During Maximum Contraction in Combat Athletes
Brief Title: Effect of Dehydration on Sleep Quality, Cognitive Skills, and Electromyographic Responses in Combat Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BAIBU-SBF-UK-03
Record Dates: First submitted 2025-07-29; First posted 2025-08-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Dehydration; Weight Loss; Weight Cycling; Sleep
Keywords: Athletic Performance; Cognitive Skills; Sleep Quality; Isokinetic strength; EMG Response; Anticipation Time
MeSH Terms: conditions — Dehydration; Weight Loss; Weight Cycling; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized counterbalanced crossover design study (Two experimental trial a control trial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dehydration + Dehydrated Night Trial (Experimental): In this trial 3% weight loss will be achieved with sauna application by taking the body weights recorded in the pre-test as a reference. Following the dehydration application, all measurements taken in the pre-test before the application will be repeated in order after approximately 45 minutes.
  Athletes will be permitted to engage in a routine night without rehydration. During this period, their sleep quality will be recorded with a sleep tracker. The next day in the morning, all measurements taken in the pre-test will be repeated in order to evaluate the effect of dehydration and the possible negative effect of dehydration on sleep quality on the dependent variables. Following the completion of the morning measurements, the athletes will be permitted to consume fluids and food within two hours in order to reach their body weights in the pre-test. All tests will be reapplied for the last time to the athletes who have reached the state of rehydration, respectively.
  Interventions: Other: Rapid weight loss through dehydration
- Dehydration + Rehydrated Night Trial (Experimental): In this trial 3% weight loss will be achieved with sauna application by taking the body weights recorded in the pre-test as a reference. Following the dehydration application, all measurements taken in the pre-test before the application will be repeated in order after approximately 45 minutes, with the athlete refraining from consuming any food or liquid. Athletes will be permitted to rehydrate after the second measurements and will be asked to spend a routine night. The remaining tests will be repeated in accordance with the experimental trial 1 protocol.
  Interventions: Other: Rapid weight loss through dehydration
- Control Trial (No Intervention): No intervention will be conducted. All tests to be used to measure dependent variables will be conducted in accordance with the Experimental trial 1 protocol.

INTERVENTIONS:
Other: Rapid weight loss through dehydration — Dehydration will be induced by exposing athletes to sauna heat with an average temperature of 70-80°C. The participants will undergo consecutive 15 minute sessions in sauna with 5 minute breaks until 3% weight loss is achieved. No liquids or food will be consumed between sessions.
  Arms: Dehydration + Dehydrated Night Trial; Dehydration + Rehydrated Night Trial

SUMMARY:
This study examines the effects of rapid dehydration-induced weight loss on combat athletes' sleep quality, cognitive skills, and isokinetic strength performance. The research documents both benefits and risks of weight-cutting practices for athletes, coaches, and medical staff in weight-class sports. Findings will guide safer weight management approaches and inform potential revisions to international weigh-in protocols, while contributing valuable insights to sports science.

DETAILED DESCRIPTION:
The objective of this study is to examine the impact of rapid weight loss through dehydration on sleep quality, cognitive skills, and surface electromyographic (sEMG) responses during isokinetic strength performance in combat athletes. Additionally, the overall effect of acute dehydration and the potential adverse effects of dehydration on sleep quality on cognitive abilities, and sEMG responses will be evaluated. Body temperature and heart rate values will be monitored throughout the study. Finally, the effect of rehydration on cognitive skills, strength, and sEMG responses after a night of dehydration will be evaluated.

Competitive senior male combat athletes will participate in this study. The first stage will involve the determination of urine density, the recording of body weight, the measurement of body composition and total body fluid, and the recording of resting heart rate (HR) and body temperature. Subsequently, cognitive skill tests will be administered, and following a standard warm-up, sEMG data will be recorded from the dominant leg quadriceps muscle region during isokinetic leg strength measurements.

Following the completion of the pre-tests, each athlete will be subjected to two separate dehydration and control applications in accordance with the randomised crossover experimental design. In the experimental trials, 3% weight loss will be achieved with sauna application by taking the body weights recorded in the pre-test as a reference. Following the dehydration application, all measurements taken in the pre-test before the application will be repeated in order after approximately 45 minutes, with the athlete refraining from consuming any food or liquid.

Athletes in experimental trial 1 will be permitted to engage in a routine night without rehydration. During this period, their sleep quality will be recorded with a sleep monitor. The next day in the morning, all measurements taken in the pre-test will be repeated in order to evaluate the effect of dehydration and the possible negative effect of dehydration on sleep quality on the dependent variables. Following the completion of the morning measurements, the athletes will be permitted to consume fluids and food within two hours in order to reach their body weights in the pre-test. All tests will be reapplied for the last time to the athletes who have reached the state of rehydration, respectively. In the experimental trial 2, they will be permitted to rehydrate after the second measurements and will be asked to spend a routine night. The remaining tests will be repeated in accordance with the experimental trial 1 protocol. In the control trial, all tests in the experimental trials will be performed without body weight loss due to dehydration. All participants will be randomly assigned to the dehydration and control trials, with each athlete participating in the respective trial at one-week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Being combat athletes with prior rapid weight loss experience
* No existing health conditions
* No orthopedic injuries

Exclusion Criteria:

* Using of sleep-related medications
* Complications During the Intervention: Participants who experience any complications during experimental intervention.

Ages: 17 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male individuals will be included due to the fact that women's hormonal responses may cause heterogeneous findings and the difficulty in interpreting the findings due to their hormonal profile.
Enrollment: 12 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep monitoring and Evaluation | First trial monitoring, following one week Second trial monitoring and following one week Third trial monitoring (Due to randomized counterbalanced crossover design, monitoring will be performed three times, two as experimental and one as control).
  Participants' sleep assessments will be conducted with a sleep monitor, which uses impulse radio ultra-wide band (IR-UWB) radar and Doppler technology, and has been shown to provide measurements as accurate and reliable as the polysomnography device, which is considered the gold standard in sleep assessment. Total sleep and wake times and durations of the sleep phases will be obtained in minutes from the recordings of the device.
Isokinetic Leg Strength Measurement | First trial testing, following one week Second trial testing and following one week Third trial testing (Due to randomized counterbalanced crossover design, testing will be performed three times, two as experimental and one as control).
  Isokinetic leg strength measurements will be made with the Cybex Norm device. Peak torque data obtained during the measurements will be recorded and used in data processing.
EMG Measurements | First trial testing, following one week Second trial testing and following one week Third trial testing (Due to randomized counterbalanced crossover design, testing will be performed three times, two as experimental and one as control).
  Electrical potentials of muscle cells are recorded with electromyography (EMG) and the activities of skeletal muscles are evaluated based on changes in these potentials. EMG measurement provides information about the muscles and motor nerves involved by analyzing motor unit action potentials.
Stroop test | First trial testing, following one week Second trial testing and following one week Third trial testing (Due to randomized counterbalanced crossover design, testing will be performed three times, two as experimental and one as control).
  The Stroop test is a test that reflects frontal lobe region activity.
Symbol Digit Modalities Test | First trial testing, following one week Second trial testing and following one week Third trial testing (Due to randomized counterbalanced crossover design, testing will be performed three times, two as experimental and one as control).
  The Symbol Digit Modalities Test is a test that evaluates complex visual spatial scanning, sustained attention and concentration, information processing speed and working memory.
Montreal Cognitive Assessment | First trial testing, following one week Second trial testing and following one week Third trial testing (Due to randomized counterbalanced crossover design, testing will be performed three times, two as experimental and one as control).
  The Montreal Cognitive Assessment test evaluates cognitive functions such as attention and concentration, executive functions, memory, language, visual construction skills, calculation and orientation. The test scores range from 0 to 30, with a cut-off score of 21. Scores of 21 and above are considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Umid Karli, PhD, Principal Investigator — Bolu Abant İzzet Baysal University, Faculty of Sport Sciences, Department of Coaching Education
Locations (1):
- Bolu Abant İzzet Baysal University, Faculty of Sport Sciences,, Bolu, Turkey (Türkiye)